CLINICAL TRIAL: NCT06246851
Title: A Clinical Study Comparing the Immune Response to Revaccination With Intradermal BCG and Aerosol BCG in Previously BCG Vaccinated Healthy Adult Volunteers With and Without Type 2 Diabetes
Brief Title: BCG Revaccination Study in Diabetic and Non-Diabetic Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TB046
Record Dates: First submitted 2023-12-19; First posted 2024-02-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: This is a phase 1 study exploring differences between the immunological responses to revaccination with intradermal-BCG and aerosol-inhaled BCG in healthy adults and those with pre-existing T2DM.
  There will be three study groups with twelve volunteers in each group. Volunteers will be enrolled into groups based upon whether they have a diagnosis of T2DM. They will then be vaccinated with intradermal BCG (Groups A and C) or aerosolised BCG (Group B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: A1: 2-8 x 10^5 cfu or 1 x 10^5 cfu intradermal BCG (non-type 2 diabetic group) (Experimental): A1: 6 historically BCG-vaccinated volunteers without type 2 diabetes will receive 2-8 X 10^5 cfu intradermally injected BCG.
  A2: 6 historically BCG-vaccinated volunteers without type 2 diabetes will receive 1 x 10^5 cfu intradermally injected BCG.
  All Group A volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish
- Group B: 2-8 x 10^6 cfu or 1 x 10^6 cfu aerosol inhaled BCG (non-type 2 diabetic group) (Experimental): B1: 6 historically BCG-vaccinated volunteers without type 2 diabetes will receive 2-8 X 10^6 cfu aerosol inhaled BCG.
  B2: 6 historically BCG-vaccinated volunteers without type 2 diabetes will receive 1 X 10^6 cfu aerosol inhaled BCG.
  All Group B volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish
- Group C: 2-8 x 10^5 cfu or 1 x 10^5 cfu intradermal BCG (type 2 diabetic group) (Experimental): C1: 6 historically BCG-vaccinated volunteers with confirmed type 2 diabetes will receive 2-8 X 10^5 cfu intradermally injected BCG.
  C2: 6 historically BCG-vaccinated volunteers with confirmed type 2 diabetes will receive 1 X 10^5 cfu intradermally injected BCG.
  All Group C volunteers will not have a bronchoscopy.
  Interventions: Biological: BCG Danish

INTERVENTIONS:
Biological: BCG Danish — BCG Danish 1331 is on the WHO list of pre-qualified vaccines and has a well-defined side effect profile. BCG is licensed for delivery via the intradermal route. It is not licensed for delivery via the aerosol route.

SUMMARY:
The purpose of this study is to:

1. explore whether investigators can make BCG more effective by giving it in a different way. For this, aerosol inhaled BCG will be compared against the conventional BCG injection.
2. explore if there are differences in response to re-vaccination in healthy volunteers with and without Type 2 Diabetes.

It will involve 36 previously BCG-vaccinated participants. Bronchoscopies will be performed 14 days post-challenge to measure BCG recovered from bronchial samples. Blood tests will be taken to look at potential immunological markers of immunity.

DETAILED DESCRIPTION:
Worldwide Tuberculosis (TB) remains the leading cause of death from an infectious disease. Key research priorities include the development of effective vaccine strategies.

Currently, the only licensed vaccine against TB is BCG (Bacille Calmette-Guérin) injected under the skin (intradermal). This works well as a single dose vaccination against TB in childhood but is often ineffective in adults. Previous studies have investigated the benefit of booster doses of intradermal BCG; although these have not shown a clear benefit in reducing the risk of getting a TB infection there is emerging evidence that it may reduce its duration. Certain groups of people are at a higher risk of infection with Mycobacterium tuberculosis, the bacterium that causes TB. An important risk group are those with Diabetes Mellitus, who are at an increased risk of both becoming infected and dying from the disease. The reason for this is not clear, however differences in the immune response to Mycobacteria are thought to be important. Strategies to improve protection of high risk groups including those with Diabetes are needed to reduce the global burden of TB.

Localised immune responses can differ to those seen systemically. Vaccine studies in other infectious diseases have shown that altering the route of administration can improve protection from disease. There is also evidence from animal studies that breathing in BCG as a fine mist (aerosol) can make the vaccine more effective than BCG injections. Previous clinical trials in our group (TB041 and TB044) and a current study (TB043) recruited healthy volunteers and showed that aerosol inhaled BCG can be safely administered. It has also been shown that BCG given this way can elicit immunological responses not seen in the systemic blood compartment. Vaccination with BCG through the respiratory tract therefore offers an important alternative to intradermal vaccination, which has the potential to be a more effective route for a boosting vaccine.

This study will provide data on the immune response to booster vaccination with BCG. The investigators will compare how these responses differ between routes of vaccine delivery (aerosol inhaled BCG versus intradermal vaccination), and also explore how the immune response to revaccination differs in adults with Type 2 diabetes (T2DM). The investigators will use the findings to explore the potential benefits of aerosol vaccination and to investigate differences in the immune responses in diabetic individuals to understand how the investigators can improve protection against TB in this high risk group.

It will involve a total of 36 previously BCG-vaccinated participants; 12 healthy volunteers will receive boosting vaccination with aerosol BCG, while a further 12 healthy volunteers will receive a boosting vaccination with intradermal BCG. The investigators will perform washings from the lungs (bronchoscopies) 14 days after BCG vaccination to measure immunological and bacterial responses. A further 12 previously BCG-vaccinated, healthy adult volunteers with T2DM will receive a boosting vaccination with intradermal BCG. The investigators will take blood samples from all volunteers to explore the immune response to BCG and to develop markers to understand who has developed a protective immune response to TB.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-65 years
* Resident in or near Oxford for the duration of the study period
* Provide written informed consent
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner (or review summary care record, if available)
* Allow the investigator to register volunteer details with a confidential database (The Over- volunteering Protection Service) to prevent concurrent entry into clinical studies/trials
* Agreement to refrain from blood donation during the course of the study
* For persons of child-bearing potential (POCBP) only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening, vaccination and bronchoscopy
* Able and willing (in the investigator's opinion) to comply with all study requirements
* No clinically relevant findings on physical examination
* Screening IGRA negative
* Willing to be tested for evidence of SARS-CoV-2 infection and to allow public health notification of the results if required
* Previously vaccinated with the BCG (at least 12 months prior to enrolment, as evidenced by a visible scar or documentation in medical or occupational health records)
* Group C only - Documented diagnosis of T2DM (made at least 12 months prior to enrolment) initiated on a management plan with medication including use of metformin

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment or during the trial follow up period
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study agent, any essential study procedure, sedative drugs, or any local or general anaesthetic agents
* Clinically significant history of skin disorder, allergy, atopy, cancer (except BCC of the skin or CIS of the cervix), bleeding disorder, cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder (excluding T2DM in Group C only), neurological illness, psychiatric disorder, drug or alcohol abuse
* Any significant autoimmune conditions or immunodeficiency (including HIV)
* Previous diagnosis or treatment for TB disease or latent TB infections
* Clinical, radiological, or laboratory evidence of current active TB disease or latent TB infection
* Previous receipt of any investigational TB vaccine or aerosolised BCG
* More than one previous BCG vaccination
* Positive HBsAg, HCV or HIV antibodies
* Concurrent use of oral, inhaled or systemic steroid medication or use for more than 14 days within the last 6 months (steroids used as a cream or ointment are permissible), or the use of other immunosuppressive agents concurrently or for more than 14 days within the last 6 months
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned study vaccination date
* Administration of a live vaccine within the preceding 28 days prior to enrolment
* Administration of any other non-live vaccine within the preceding 14 days prior to enrolment
* Pregnancy, lactation or intention to become pregnant during study period
* Previously resident for more than 12 months concurrently in the rural areas of a tropical climate where significant non-tuberculous mycobacterial exposure is likely
* Any other clinically significant abnormality of screening blood or urine tests
* Any other significant disease, disorder, or finding, which, in the opinion of the investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data
* A body mass index (BMI) of <18.5 or >45

Group A or B Specific Exclusions:

* Any clinically significant respiratory disease, including asthma
* Current smoker (defined as any smoking including e-cigarettes in the last 3 months)
* Current use of any medication or other drug taken through the nasal or inhaled route including cocaine or other recreational drugs
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Shares a household with someone with clinically significant immunodeficiency (either from infection or medication) who is deemed to be at risk of developing disseminated BCG infection if exposed to BCG
* An HBA1c at screening of > 48mmol/Lmol
* Clinically significant abnormality on screening chest radiograph
* Clinically significant abnormality of lung function testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Intradermal vs. aerosol BCG in non-type 2 diabetics | Up to day 168
  To compare the immunological response of BCG re-vaccination by the aerosol inhaled route to the intradermal route in healthy historically intradermally BCG-vaccinated volunteers.
  This will be measured using laboratory markers of innate and adaptive immunity, which may include ex-vivo ELISpot and ELISAs, RNA sequence analysis and intracellular cytokine staining of blood. This will also be measured using flow cytometry, ELISA and cytokine staining of BAL samples.
  This will be achieved by blood test done at each follow up visit and bronchoscopy to retrieve BAL sample at Day 14 visit for non- diabetic volunteers.
Intradermal (in type 2 diabetics) vs intradermal (in non-type 2 diabetics) | Up to day 168
  To compare the immunological response of BCG re-vaccination by the intradermal route in historically intradermally BCG-vaccinated volunteers with Type 2 Diabetes and non-diabetic healthy adults.
  This will be measured using laboratory markers of innate and adaptive immunity, which may include ex-vivo ELISPOT and ELISAs, RNA sequence analysis and intracellular cytokine staining of blood.
  This will be achieved through the blood test done at each follow up visit.

SECONDARY OUTCOMES:
Intradermal or aerosol BCG re-vaccination safety in healthy volunteers | Up to day 168
  To describe the safety of intradermal or aerosol BCG as a BCG re-vaccination in healthy UK Volunteers.
  This will be measured using actively and passively collected data on adverse events and detailed participant symptom profiles throughout the study duration.

OTHER OUTCOMES:
Examination of immunological and microbiological markers | Up to day 168
  To examine immunological and microbiological markers that correlate with increased protection from M.tb infection.
  This will be measured using laboratory markers of innate and adaptive immunity, which may include the Mycobacterial Growth Inhibition assay on PBMC/serum and on BAL cells, ex-vivo ELISpot and ELISAs, RNA sequence analysis and intracellular cytokine staining of blood. This will also be measured using flow cytometry, ELISA, cytokine staining and other exploratory immunology or microbiology assays on blood or respiratory samples.
  This will be achieved through blood test and swabs at each follow up visits and bronchoscopy at Day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Professor, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom